CLINICAL TRIAL: NCT02287025
Title: Does Physician Education Influence Side Effect Management and Does it Increase Time on Treatment in the Absence of Progression ? A Phase 4 Open-label Trial With Regorafenib in Metastatic Colorectal Cancer
Brief Title: A Phase 4 Study of Regorafenib in Metastatic Colorectal Cancer - Does Educating Physicians Change Patient Outcomes?
Acronym: SMART
Status: Terminated | Phase: Phase 4 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 17347
Record Dates: First submitted 2014-10-07; First posted 2014-11-10 (Estimated); Results first posted 2017-10-19 (Actual); Last update posted 2017-10-19 (Actual); Status verified 2017-07

CONDITIONS: Physician Education
MeSH Terms: interventions — regorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- SMART (Experimental): Investigators were supported with enhanced drug-specific information via an iPad application (SMART).
  Interventions: Drug: Regorafenib (Stivarga, BAY73-4506); Other: iPAD application
- Standard of Care (Active Comparator): Investigators were supported with standard prescribing information.
  Interventions: Drug: Regorafenib (Stivarga, BAY73-4506); Other: Bayer specialist

INTERVENTIONS:
Drug: Regorafenib (Stivarga, BAY73-4506) — Dose(s) 160 mg tablet (4 tablets per day at 40 mg) daily for 3 weeks on / 1 week off
Other: iPAD application — Investigators were supported with enhanced drug-specific information via an iPad application (SMART).
  Arms: SMART
Other: Bayer specialist — The treating investigator will have access to the prescribing information and have ability to consult a Bayer specialist, should questions arise.
  Arms: Standard of Care

SUMMARY:
Randomized trial to evaluate impact of healthcare provider( clinician and nursing staff) support and education on treatment discontinuation rates in the absence of progression in patients with metastatic colorectal cancer treated with regorafenib. Intensified education and support will be provided through an application for iPad which has automatic links to grading, dose reduction and side effect management ,as well as, references for additional articles.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically-proven metastatic CRC for which the decision of treatment with regorafenib was made
* Previous treatment with fluoropyrimidine-, oxaliplatin- and irinotecan-based chemotherapy, an anti-VEGF therapy, and, if KRAS wild type, an anti-EGFR therapy
* Male or female patients ≥ 18 years of age
* Eastern Cooperative Oncology Group performance status (ECOG PS) of 0 or 1
* Signed informed consent obtained before any study specific procedure is performed.Patients must be able to understand and willing to sign the written ICF.
* Life expectancy of at least 12 weeks
* Adequate bone marrow, liver and renal function as assessed by the following laboratory requirements:

  1. Total bilirubin ≤ 1.5 x the upper limits of normal (ULN)
  2. Alanine aminotransferase (ALT) and aspartate aminotransferease (AST)

     ≤ 3.0 x ULN (≤ 5 x ULN for patients with liver involvement of their cancer)
  3. Alkaline phosphastase limit ≤ 2.5 x ULN (≤ 5 x ULN for patients with liver involvement of their cancer)
  4. Lipase ≤ 1.5 x the ULN
  5. Amylase ≤ 1.5 x the ULN
  6. Serum creatinine ≤ 1.5 x the ULN
  7. International normalized ratio (INR) ≤ 1.5 x ULN and partial thromboplastin time (PTT) or activated partial thromboplastin time (aPTT) ≤ 1.5 x ULN unless receiving treatment with therapeutic anticoagulation. Patients being treated with anticoagulant (e.g., heparin), will be allowed to participate provided no prior evidence of an underlying abnormality in these parameters exists. Close monitoring of at least weekly evaluations will be performed until INR and PTT are stable based on a pre-dose measurement as defined by the local standard of care.
  8. Platelet count ≥ 100000 /mm3, hemoglobin (Hb) ≥ 9 g/dL, absolute neutrophil count (ANC) ≥ 1500/mm3. Blood transfusion to meet the inclusion criteria will not be allowed.
* Estimated creatinine clearance (CLcr) ≥ 30 mL/min as calculated using the Cockroft-Gault (C-G) equation.
* Women of childbearing potential must have a blood or urine pregnancy test performed a maximum of 7 days before start of study treatment, and a negative result must be documented before start of study treatment.
* Women of childbearing potential and men must agree to use adequate contraception before entering the program until at least 8 weeks after the last study drug administration.

Exclusion Criteria:

* Unable to swallow oral medications.
* Prior use of regorafenib
* Previous assignment to treatment during this study. Patients permanently withdrawn from study participation will not be allowed to re-enter study.
* Uncontrolled hypertension (systolic blood pressure > 140 millimeters of mercury (mmHg) or diastolic pressure > 90 mmHg despite optimal medical management)
* Active or clinically significant cardiac disease including:

  1. Congestive heart failure - New York Heart Association (NYHA) > Class II
  2. Active coronary artery disease
  3. Cardiac arrhythmias requiring anti-arrhythmic therapy other than beta blockers or digoxin
  4. Unstable angina (anginal symptoms at rest), new-onset angina within 3 months before randomization, or myocardial infarction within 6 months before randomization
* Evidence or history of bleeding diathesis or coagulopathy, irrespective of severity
* Any hemorrhage or bleeding event > National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) Grade 3 within 4 weeks prior to the start of study medication
* Arterial or venous thrombotic or embolic events such as cerebrovascular accident (including transient ischemic attacks), deep vein thrombosis or pulmonary embolism within 6 month before the start of study medication (except for adequately treated catheter-related venous thrombosis occurring more than one month before the start of study medication)
* Previously untreated or concurrent cancer that is distinct in primary site or histology from colorectal cancer except cervical cancer in-situ, treated basal cell carcinoma, or superficial bladder tumor. Patients surviving a cancer that was curatively treated and without evidence of disease for more than 3 years before randomization are allowed.All cancer treatments must be completed at least 3 years prior to study entry (i.e.,signature date of the ICF).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2014-11-11 (Actual); Primary Completion 2016-02-26 (Actual); Study Completion 2016-04-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (16):
- United States (16):
  - Anniston, Alabama
  - Anaheim, California
  - Orange, California
  - Lake City, Florida
  - Skokie, Illinois
  - Lafayette, Indiana
  - Columbia, Maryland
  - Fayetteville, North Carolina
  - Canton, Ohio
  - Tulsa, Oklahoma
  - Gettysburg, Pennsylvania
  - Kingsport, Tennessee
  - Houston, Texas
  - Tyler, Texas
  - Bristol, Virginia
  - Portsmouth, Virginia

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 10 study centers in United States, from 11 NOV 2014 (first subject first visit) to 26 FEB 2016 (last subject last visit).
Pre-assignment Details: Of the 23 screen participants, 2 participants were screen fails, 2 consented but never started treatment due to early study termination and 19 patients entered treatment.
Units Other Than Participants: study sites
Period: Overall Study
Arm/Group | SMART | Standard of Care
Started | 12; 6 study sites | 11; 4 study sites
Completed | 2; 6 study sites | 2; 4 study sites
Not Completed | 10; 0 study sites | 9; 0 study sites
Not completed — Not treated | 2 | 0
Not completed — Progression of disease | 3 | 2
Not completed — Adverse Event | 2 | 4
Not completed — Withdrawal by Subject | 2 | 2
Not completed — Screening failed | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- SMART: Participants received 160 mg tablet (4 tablets per day at 40 mg) daily for 3 weeks on / 1 week off. Investigators were supported with enhanced drug-specific information via an iPad application (SMART).
- Standard of Care: Participants received 160 mg tablet (4 tablets per day at 40 mg) daily for 3 weeks on / 1 week off. Investigators were supported with standard prescribing information.
- Total: Total of all reporting groups
Arm/Group | SMART | Standard of Care | Total
Number analyzed (Participants) | 12 | 11 | 23
Age, Continuous [Mean (Standard Deviation); unit: Years] | 61.08 (15.28) | 59.91 (4.29) | 60.52 (11.70)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 3 | 9
  Male | 6 | 8 | 14

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Patients Who Discontinue Prior to Documented Progression of Disease (PD) or Death
Time Frame: Up to 1 year
Population: The study was pre-maturely terminated. No data were collected from participants for this assessment.
Groups:
- Regorafenib (Stivarga, BAY 73-4506): Dose(s) 160 mg tablet (4 tablets per day at 40 mg) daily for 3 weeks on / 1 week off
Arm/Group | Regorafenib (Stivarga, BAY 73-4506)
Number analyzed (Participants) | 0

2. Secondary Outcome: Duration of Treatment
Time Frame: Up to 1 year
Population: The study was pre-maturely terminated. No data were collected from participants for this assessment.
Arm/Group | Regorafenib (Stivarga, BAY 73-4506)
Number analyzed (Participants) | 0

3. Secondary Outcome: Dose Intensity as Percentage of Planned Dose
Description: Dose level 0 (standard starting dose) @ 160mg po qd. Dose level - 1 @ 120 mg po qd. Dose level - 2 @ 80 mg po qd. This schedule reflects the FDA-approved dosing specified in the prescribing information.
Time Frame: Up to 1 year
Population: The study was pre-maturely terminated. No data were collected from participants for this assessment.
Arm/Group | Regorafenib (Stivarga, BAY 73-4506)
Number analyzed (Participants) | 0

4. Secondary Outcome: Incidence of Grade 3 Hand-foot-skin Reaction (HFSR), Fatigue, Diarrhea, Hypertension
Description: Documented during visits as part of the interval history. All AEs will be reported in the CRF with a diagnosis, start/stop dates, action taken.
Time Frame: Up to 1 year
Population: The study was pre-maturely terminated. No data were collected from participants for this assessment.
Arm/Group | Regorafenib (Stivarga, BAY 73-4506)
Number analyzed (Participants) | 0

5. Secondary Outcome: Investigator Comfort With the Use of Regorafenib and Management of AEs as Measured by Questionnaire
Description: Investigator comfort of managing adverse events, adjusting dosing schedule, and satisfaction with SMART application measured by a questionnaire; 10 categories were answered on a 1 - 7 scale.
Time Frame: Up to 1 year
Population: The study was pre-maturely terminated. No data were collected from participants for this assessment.
Arm/Group | Regorafenib (Stivarga, BAY 73-4506)
Number analyzed (Participants) | 0

6. Secondary Outcome: Satisfaction of Investigator/Nurse With Enhanced Drug-specific Information Via SMART Questionnaire
Description: as for outcome 5
Time Frame: Up to 1 year
Population: The study was pre-maturely terminated. No data were collected from participants for this assessment.
Arm/Group | Regorafenib (Stivarga, BAY 73-4506)
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: All AEs occurring from the time the subject has signed ICF until 30 days after the last dose of study drug
Description: SAF (N= 19) included all subjects who received at least one dose of the study medication.
Arm/Group | Regorafenib (Stivarga, BAY 73-4506)
Serious Adverse Events (participants affected / at risk) | 3/19
Other Adverse Events (participants affected / at risk) | 18/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Regorafenib (Stivarga, BAY 73-4506) (N=19)
HEART FAILURE (Cardiac disorders) | 1 (1)
FEVER (General disorders) | 1 (1)
HEPATIC FAILURE (Hepatobiliary disorders) | 1 (1)
PNEUMONIA (Infections and infestations) | 1 (1)
HEMORRHAGE BRAIN (Nervous system disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Regorafenib (Stivarga, BAY 73-4506) (N=19)
ANEMIA (Blood and lymphatic system disorders) | 1 (1)
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 2 (5)
HYPOTHYROIDISM (Endocrine disorders) | 1 (1)
BLURRED VISION (Eye disorders) | 1 (2)
CONJUNCTIVITIS (Eye disorders) | 1 (1)
ABDOMINAL PAIN (Gastrointestinal disorders) | 6 (7)
CONSTIPATION (Gastrointestinal disorders) | 7 (8)
DIARRHEA (Gastrointestinal disorders) | 9 (21)
DRY MOUTH (Gastrointestinal disorders) | 2 (2)
DYSPHAGIA (Gastrointestinal disorders) | 1 (1)
FLATULENCE (Gastrointestinal disorders) | 1 (1)
GASTROESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 1 (1)
LIP SWELLING (Gastrointestinal disorders) | 1 (2)
NAUSEA (Gastrointestinal disorders) | 7 (8)
OROPHARYNGEAL CONDITIONS (Gastrointestinal disorders) | 1 (1)
PROCTITIS (Gastrointestinal disorders) | 1 (2)
SORES MOUTH (Gastrointestinal disorders) | 2 (2)
STOOL DISCOLORED (Gastrointestinal disorders) | 1 (1)
VOMITING (Gastrointestinal disorders) | 5 (6)
ASTHENIA (General disorders) | 2 (2)
CHEST PAIN (General disorders) | 1 (1)
CHILLS (General disorders) | 1 (1)
FATIGUE (General disorders) | 12 (18)
FEVER (General disorders) | 4 (5)
GAIT DISTURBANCE (General disorders) | 1 (1)
OEDEMA PERIPHERAL (General disorders) | 1 (1)
PAIN (General disorders) | 1 (1)
PERIPHERAL SWELLING (General disorders) | 1 (1)
RASH GENERALIZED (General disorders) | 1 (1)
SLIGHT FEVER (General disorders) | 1 (1)
SWELLING OF LEGS (General disorders) | 1 (1)
ALANINE AMINOTRANSFERASE INCREASED (Hepatobiliary disorders) | 3 (3)
ALKALINE PHOSPHATASE INCREASED (Hepatobiliary disorders) | 1 (1)
ALT INCREASED (Hepatobiliary disorders) | 1 (1)
ASPARTATE AMINOTRANSFERASE INCREASED (Hepatobiliary disorders) | 1 (1)
AST INCREASED (Hepatobiliary disorders) | 1 (1)
BLOOD BILIRUBIN INCREASED (Hepatobiliary disorders) | 2 (2)
HYPERBILIRUBINEMIA (Hepatobiliary disorders) | 2 (3)
LIVER FUNCTION TEST ABNORMAL (Hepatobiliary disorders) | 1 (1)
ALLERGIC REACTION TO ANTIBIOTIC (Immune system disorders) | 2 (2)
UPPER RESPIRATORY INFECTION (Infections and infestations) | 1 (1)
URINARY TRACT INFECTION (Infections and infestations) | 1 (1)
DERMATITIS RADIATION (Injury, poisoning and procedural complications) | 1 (1)
ANOREXIA (Metabolism and nutrition disorders) | 7 (8)
DECREASED APPETITE (Metabolism and nutrition disorders) | 2 (2)
HYPERGLYCEMIA (Metabolism and nutrition disorders) | 1 (1)
HYPOCALCEMIA (Metabolism and nutrition disorders) | 1 (1)
HYPOPHOSPHATEMIA (Metabolism and nutrition disorders) | 3 (3)
WEIGHT LOSS (Metabolism and nutrition disorders) | 3 (3)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 2 (2)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 2 (3)
BILATERAL MUSCLE WEAKNESS LOWER LIMB (Musculoskeletal and connective tissue disorders) | 1 (1)
BUTTOCK PAIN (Musculoskeletal and connective tissue disorders) | 1 (1)
FOOT PAIN (Musculoskeletal and connective tissue disorders) | 2 (2)
GENERALIZED MUSCLE WEAKNESS (Musculoskeletal and connective tissue disorders) | 2 (2)
JOINT SWELLING (Musculoskeletal and connective tissue disorders) | 1 (1)
LOW BACK PAIN (Musculoskeletal and connective tissue disorders) | 2 (2)
MUSCLE SPASM (Musculoskeletal and connective tissue disorders) | 1 (3)
MYALGIA (Musculoskeletal and connective tissue disorders) | 1 (1)
NECK PAIN (Musculoskeletal and connective tissue disorders) | 1 (1)
PAIN IN BACK (Musculoskeletal and connective tissue disorders) | 1 (1)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 2 (2)
PAIN IN HIP (Musculoskeletal and connective tissue disorders) | 1 (1)
UNILATERAL LEG PAIN (Musculoskeletal and connective tissue disorders) | 2 (2)
DIZZINESS (Nervous system disorders) | 3 (4)
DYSGEUSIA (Nervous system disorders) | 2 (3)
HEADACHE (Nervous system disorders) | 6 (7)
LETHARGY (Nervous system disorders) | 1 (1)
PERIPHERAL MOTOR NEUROPATHY (Nervous system disorders) | 1 (1)
POSITIONAL LIGHTHEADEDNESS (Nervous system disorders) | 1 (1)
ANXIETY (Psychiatric disorders) | 2 (2)
DEPRESSION (Psychiatric disorders) | 1 (1)
HALLUCINATIONS (Psychiatric disorders) | 1 (1)
INSOMNIA (Psychiatric disorders) | 1 (1)
DYSURIA (Renal and urinary disorders) | 2 (2)
URINARY URGENCY (Renal and urinary disorders) | 2 (2)
URINE DISCOLORATION (Renal and urinary disorders) | 2 (2)
VAGINAL DRYNESS (Reproductive system and breast disorders) | 1 (1)
COUGH (Respiratory, thoracic and mediastinal disorders) | 1 (1)
DYSPHONIA (Respiratory, thoracic and mediastinal disorders) | 1 (1)
DYSPNEA (Respiratory, thoracic and mediastinal disorders) | 2 (2)
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 4 (4)
HEMOPTYSIS (Respiratory, thoracic and mediastinal disorders) | 1 (1)
HOARSENESS (Respiratory, thoracic and mediastinal disorders) | 4 (4)
LARYNGEAL INFLAMMATION (Respiratory, thoracic and mediastinal disorders) | 1 (1)
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 1 (1)
SHORTNESS OF BREATH (Respiratory, thoracic and mediastinal disorders) | 3 (4)
SORE THROAT (Respiratory, thoracic and mediastinal disorders) | 3 (3)
ALOPECIA (Skin and subcutaneous tissue disorders) | 3 (3)
DRY SKIN (Skin and subcutaneous tissue disorders) | 2 (2)
ECZEMA (Skin and subcutaneous tissue disorders) | 1 (1)
FLUSHING (Skin and subcutaneous tissue disorders) | 2 (2)
HAND AND FOOT REACTION (Skin and subcutaneous tissue disorders) | 2 (2)
HAND AND FOOT SYNDROME (Skin and subcutaneous tissue disorders) | 5 (10)
PALMAR-PLANTAR ERYTHRODYSESTHESIA SYNDROME (Skin and subcutaneous tissue disorders) | 1 (2)
PRURITUS (Skin and subcutaneous tissue disorders) | 2 (3)
RASH ACNEIFORM (Skin and subcutaneous tissue disorders) | 1 (1)
HEMATOMA (Vascular disorders) | 1 (1)
HYPERTENSION (Vascular disorders) | 3 (9)
HYPOTENSION (Vascular disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
The study was terminated prematurely due to slow recruitment (23/300 subjects enrolled). No statistical analyses of efficacy parameters were performed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days